CLINICAL TRIAL: NCT04015843
Title: Compliance of Blood Pressure and Lipid in Hypertensive Patients Under the Management of Hospitals at Different Levels: a Real-world Observational Study
Brief Title: Compliance of Blood Pressure and Lipid in Hypertensive Patients Under the Management of Hospitals at Different Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Cardiovascular Association (Other)
Responsible Party: Sponsor
Other Study IDs: GUSU18006
Record Dates: First submitted 2019-07-03; First posted 2019-07-11 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, prospective cohort study that collects only diagnostic and therapeutic data in subjects but does not interfere with treatment.

DETAILED DESCRIPTION:
The study aims to assess blood pressure and lipid levels, the use of lipid-lowering and antihypertensive drugs, and treatment compliance and adverse events in hypertensive outpatients of 30 hospitals of different levels, following them up for 1 and 3 months after treatment, respectively. The study would reveal the compliance of blood pressure and lipid levels in hypertensive patients under management of hospitals at different levels, and analyze factors affecting blood pressure or lipid levels associated with treatment compliance. Therefore, the study would provide clinical data from the real world for future prevention and control of CVD in China.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria will be included:

1. Age ≥18 years, male or female;
2. Agreement for blood pressure and lipid testing;
3. Initial diagnosis of primary hypertension, with blood pressure conforming to the diagnostic criteria of the 2018 Guidelines for the Prevention and Treatment of Hypertension in China [14] (with no antihypertensive drugs, SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg after three tests performed on different days); or a history of primary hypertension but incompliant blood pressure;
4. Willingness to participate in the study and signing of informed consent.

Exclusion Criteria:

* Patients meeting the following criteria will be excluded:

  1. Involvement in an interventional clinical research;
  2. Pregnancy or lactation in women;
  3. Complication with malignant tumors;
  4. Diagnosis of non-primary hypertension by researchers;
  5. Impaired cognitive ability;
  6. Researchers believing that the patients have other conditions not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initial diagnosis of primary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be compliance of blood pressure in hypertensive patients after 3 months of treatment in hospitals at different levels. | 3 months
  Blood pressure measurement:
  Blood pressure in both upper arms will be measured with a sphygmomanometer, with the patient in the sitting position. The mean value of three tests will be used for statistics. When left and right upper arms show different blood pressures, the higher value will be used for statistics.

SECONDARY OUTCOMES:
Percentage of outpatients with abnormal blood lipid levels in hospitals at different levels | 3 months
  On a CardioChek dry-type biochemical analyzer, the levels of total cholesterol (TC), triglyceride (TG), high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C) in fingertip blood samples will be measured after 12-h fasting
Achievement rate of blood lipid levels in hypertensive and dyslipidemic patients after 3 months of treatment in hospitals at different levels | 3 months
  Achievement rate of blood lipid levels in hypertensive and dyslipidemic patients after 3 months of treatment in hospitals at different levels
Compliance of patients towards antihypertensive and lipid-lowering treatments in hospitals at different levels | 3 months
  Compliance of patients towards antihypertensive and lipid-lowering treatments in hospitals at different levels
Factors affecting blood pressure and lipid compliance in different hospitals, such as patient adverse events | 3 months
  Factors affecting blood pressure and lipid compliance in different hospitals, such as patient adverse events
Achievement rate of blood pressure in hypertensive patients under different levels of hospital management after 1 month of treatment | 1 months
  Achievement rate of blood pressure in hypertensive patients under different levels of hospital management after 1 month of treatment

CONTACTS AND LOCATIONS:
Overall Officials: yong huo, master, Principal Investigator — Peking University First Hospital
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No